CLINICAL TRIAL: NCT00925886
Title: Use of Toric Intraocular Lens to Neutralize Keratometric Astigmatism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-01
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cataract; Astigmatism
Keywords: Astigmatism; Cataract
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acrysof Toric intraocular lens (Experimental): A One piece, acrylic intraocular lens is implanted in the lens bag.
  Interventions: Procedure: Acrysof Toric one-piece intraocular lens

INTERVENTIONS:
Procedure: Acrysof Toric one-piece intraocular lens — Cataract Surgery with a intraocular lens implantation
  Other Names: Acrysof Single Piece Natural Toric Lens. ALCON LABORATORIES INC

SUMMARY:
The purpose of this study is to evaluate neutralization of keratometric astigmatism in patients with cataract and astigmatism higher than 1 diopter, with phaco surgery and the implantation of a toric intraocular lens.

DETAILED DESCRIPTION:
Patients with Cataract are treated with phacoemulsification of the lens with an implantation of an intraocular lens. Besides cataract, almost 25% of these patients have some degree of Astigmatism; when it is higher than 1 diopter, it is possible to neutralize it with an implantation of a toric intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

* Symmetrical keratometric astigmatism ≥ 1.0 D and cataract.

Exclusion Criteria:

* Irregular astigmatism,
* Keratoconus,
* Previous Refractive Surgery.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Neutralization of Astigmatism | 3 months after cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Asociacion Para Evitar la Ceguera en Mexico, Mexico City, D.F., Mexico

REFERENCES:
- [Background] Bauer NJ, de Vries NE, Webers CA, Hendrikse F, Nuijts RM. Astigmatism management in cataract surgery with the AcrySof toric intraocular lens. J Cataract Refract Surg. 2008 Sep;34(9):1483-8. doi: 10.1016/j.jcrs.2008.05.031. PMID 18721707